CLINICAL TRIAL: NCT00073827
Title: An Efficacy and Safety Study of Levalbuterol, Racemic Albuterol and Placebo in Subjects Twelve Years of Age and Older With Asthma
Brief Title: Study of Levalbuterol, Racemic Albuterol and Placebo in Subjects Twelve Years of Age and Older With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 051-353
Record Dates: First submitted 2003-12-09; First posted 2003-12-11 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Asthma
Keywords: adolescent; adult; asthma; levalbuterol; bronchoconstriction
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): levalbuterol MDI 90 mcg QID
  Interventions: Drug: levalbuterol tartrate MDI
- 2 (Active Comparator): racemic albuterol MDI 180 mcg QID
  Interventions: Drug: racemic albuterol MDI
- 3 (Placebo Comparator): Placebo MDI QID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: levalbuterol tartrate MDI — levalbuterol 90 mcg QID
  Other Names: Xopenex MDI
  Arms: 1
Drug: racemic albuterol MDI — racemic albuterol 180 mcg QID
  Arms: 2
Drug: Placebo — Placebo MDI QID
  Arms: 3

SUMMARY:
The primary purpose of this study was to investigate the efficacy of levalbuterol compared to a placebo and compared to albuterol in the treatment and prevention of bronchoconstriction in adolescent and adult subjects with asthma, with all treatments administered 4 times a day (QID).

DETAILED DESCRIPTION:
This was a Phase III, multicenter, randomized, double-blind, placebo- and active-controlled, parallel-group study of up to 9 weeks in duration. Seven days of QID single-blind placebo administration (via MDI) was followed by 56 days of QID double-blind active treatment. Following the run-in period, each subject was randomized to one of the following three treatments: levalbuterol HFA MDI 90 mcg (2 actuations of 45 mcg), racemic albuterol HFA MDI 180 mcg (2 actuations of 90 mcg), or placebo (2 actuations). Subjects were randomized in a 2:1:1 ratio of levalbuterol to racemic albuterol to placebo. In order to maintain blinding of the device, a placebo dose was administered with each treatment. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria

* Willing and able to comply with the study procedures and visit schedules
* Male or female, at least 12 years of age
* Female subjects 12-60 years of age must have a negative serum pregnancy test at study start.
* Women of child bearing potential must be using an acceptable method of birth control
* Have a documented diagnosis of asthma for a minimum of 6 months prior to study start
* Must have stable baseline asthma and have been using a B-adrenergic agonist, and/or anti-asthma anti-inflammatory medication, and/or OTC asthma medication for at least 6 months prior to study start
* Must be in good health with the exception of their reversible airways disease and not suffering from any chronic condition that might affect their respiratory function
* Must have a chest X-ray that is not diagnostic of pneumonia, atelectasis, pulmonary fibrotic disease, pneumothorax, chronic obstructive pulmonary disease, etc.
* Must be able to complete the diary cards and medical event calendars reliably on a daily basis, understand dosing instructions, and demonstrate how to use the MiniWright PEF meter.

Exclusion Criteria

* Female subject who is pregnant or lactating
* Have participated in an investigational drug study within 30 days prior to study start, or who is currently participating in another clinical trial
* Subject whose schedule prevents him or her from taking the first daily dose of study medication and/or starting study visits before 9 AM
* Subject who has travel commitments during the study that would interfere with trial measurements or compliance
* Have a history of hospitalization for asthma within 45 days prior to study start, or who is scheduled for in-patient hospitalization, including elective surgery
* Have a known sensitivity to levalbuterol or racemic albuterol, or any excipients in any of these formulations
* Subject using any prescription drug with which albuterol sulfate administration is contraindicated
* Subject with currently diagnosed life-threatening asthma
* History of cancer (exception: basal cell carcinoma in remission).
* Subject with hyperthyroidism, diabetes, hypertension, cardiac diseases or seizure disorders that currently are not well controlled by medication
* History of substance abuse or drug abuse within 12 months preceding study start
* Subject with greater than 10 pack year history of cigarette smoking or use of any tobacco products within 6 months of study start
* Documented history of bronchopulmonary aspergillosis or any form of allergic alveolitis
* Have suffered from a clinically significant upper or lower respiratory tract infection in the 2 weeks prior to study start
* Subject who is a staff member or relative of a staff member

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 445 (Actual)
Dates: Start 2002-05; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
percent change in FEV1 from visit predose averaged over the 8-week double-blind period | Weeks 0, 4, 8

SECONDARY OUTCOMES:
area under the FEV1 percent change curve from visit pre-dose and from study baseline curves averaged over the double-blind period | Weeks 0, 4, 8
peak percent change in FEV1 from study baseline | Weeks 0, 4, 8
peak change in FEV1 from visit predose | Weeks 0, 4, 8
peak percent of predicted FEV1 | Weeks 0, 4, 8
area under the FEV1 curve (AUC) | Weeks 0, 4, 8
peak change and peak percent change in FEF25-75% from visit predose | Weeks 0, 4, 8
peak change and peak percent change in FVC from visit predose | Weeks 0, 4, 8

CONTACTS AND LOCATIONS:
Locations (63):
- United States (63):
  - Alabama Asthma and Allergy Center, Homewood, Alabama
  - MDC Research, Mobile, Alabama
  - Integrated Research Group, Corona, California
  - Allergy & Asthma Medical Group of Diablo Valley, Inc., Danville, California
  - Radiant Research, Inc., Encinitas, California
  - Allergy & Asthma Specialists Medical Group, Huntington Beach, California
  - Allergy, Asthma & Respiratory Care Center, Long Beach, California
  - Allergy Research Foundation, Inc., Los Angeles, California
  - Clinical Trials of Orange County, Orange, California
  - Allergy Associates Medical Group, San Diego, California
  - Allergy & Asthma Medical Group & Research Center, San Diego, California
  - Allergy & Asthma Prevention & Treatment Center, San Diego, California
  - Allergy & Asthma Assoc. of Santa Clara Valley Research Center, San Jose, California
  - Bensch Research Associates, Stockton, California
  - Southern California Research Center, Viejo, California
  - National Jewish Medical & Research Center, Denver, Colorado
  - Clinical Research Centers of Colorado PC, Englewood, Colorado
  - Asthma & Allergy Associates, PC, Pueblo, Colorado
  - Office of Ronald Saff, Tallahassee, Florida
  - Aeroallergy Research Laboratories of Savannah, Inc., Savannah, Georgia
  - Radiant Research Honolulu, Honolulu, Hawaii
  - Clinical Research Center of Indiana, Indianapolis, Indiana
  - Allergy & Asthma Care Specialists, Metairie, Louisiana
  - Northshore Medical Research, Slidell, Louisiana
  - University of Maryland School of Medicine, Baltimore, Maryland
  - PCHI, Needham, Massachusetts
  - Northeast Medical Research Associates, Inc., North Dartmouth, Massachusetts
  - Center for Clinical Research, Taunton, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Clinical Research Institute, Minneapolis, Minnesota
  - Mississippi Asthma & Allergy Clinic, Jackson, Mississippi
  - Office of Clinical Research, University of Missouri-Columbia, Columbia, Missouri
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Division of Allergy & Immunology, Washington Univ School of Med, St Louis, Missouri
  - St. Louis University, St Louis, Missouri
  - The Clinical Research Center, LLC, St Louis, Missouri
  - Princeton Center for Clinical Research, Princeton, New Jersey
  - Pulmonary and Allergy Associates, Springfield, New Jersey
  - PCCS, Albany, New York
  - AAIR Research Center, Rochester, New York
  - Regional Allergy & Asthma Consultants, Asheville, North Carolina
  - Cornerstone Research Care, High Point, North Carolina
  - Raleigh Pediatric Associates, Raleigh, North Carolina
  - Bernstein Clinical Research Center, LLC, Cincinnati, Ohio
  - Allergy & Asthma Research, Eugene, Oregon
  - Allergy Associates Research Center, LLC, Portland, Oregon
  - Asthma & Allergy Research Associates, Chester, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh Division of Allergy, Immunology & Infectious Diseases, Pittsburgh, Pennsylvania
  - University of Pittsburgh Division of Pulmonary, Pittsburgh, Pennsylvania
  - Radiant Research, Charleston, South Carolina
  - Office of Neil Kao, Greenville, South Carolina
  - Allergy & Asthma Consultants, LLP, Mt. Pleasant, South Carolina
  - Office of Constantine Saadeh, Amarillo, Texas
  - Allergy & Asthma Research Associates, Dallas, Texas
  - North Texas Institute for Clinical Trials, Fort Worth, Texas
  - Breath of Life Research Institute, Houston, Texas
  - Lung Diagnostics, San Antonio, Texas
  - Allergy & Asthma Center, Waco, Texas
  - Children's Hospital of the Kings Daughters, Norfolk, Virginia
  - Pulmonary Associates of Richmond, Inc., Richmond, Virginia
  - ASTHMA, Inc., Seattle, Washington
  - Allergic Diseases, SC, West Allis, Wisconsin